CLINICAL TRIAL: NCT02022319
Title: Intra- and Inter-observer Variation of Thyroid Shear Wave Elastography - a Variability Study
Brief Title: The Observer Variation of Shear Wave Elastography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristine Zøylner Rubeck, MD, University of Aarhus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SWE-var 112013
Record Dates: First submitted 2013-12-15; First posted 2013-12-27 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Thyroid Nodular Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Shear Wave Elastography (Other): All included patients undergo a supplementary Shear Wave Elastographic scan
  Interventions: Device: Ultrasonographic Shear Wave Elastography

INTERVENTIONS:
Device: Ultrasonographic Shear Wave Elastography

SUMMARY:
Background: The main goal of diagnosing thyroid nodules is to differentiate the few malignant from the large background of benign lesion. Currently available pre-operative tests are unable to rule out malignancy in a subset of patients and diagnostic surgery is necessary. Therefore there is a need to develope the available diagnostic tools for the pre-operative diagnostic work-up of thyroid nodules.

The study will investigate a novel ultrasonographic technique called Shear Wave Elastography (SWE) in the pre-operative evaluation of thyroid nodules.

Hypothesis:

1) SWE is a precise tool for evaluation of thyroid nodules in terms of inter- and intra-observer reliability and day-to-day variation.

The study will be conducted as part of a larger PhD study, and an evaluation of the diagnostic value of thyroid SWE will be evaluated in a larger study.

Perspectives:

An optimization of the pre-operative risk-stratification and diagnosis of thyroid nodules can reduce unnecessary thyroid surgery, with a reduction in morbidity and better use of the economic and surgical resources.

ELIGIBILITY:
Inclusion Criteria:

* patients with a thyroid nodule ≥1 cm in largest dimension (solitary or dominating nodule in multinodular goiter),
* Patients undergoing thyroid surgery.

Exclusion Criteria:

* Nodules located in the isthmus of the thyroid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Elasticity index | Repeat measures obtained on the same day (ten minutes to one hour between measurements), and measures obtained on a different day (one day to several weeks).
  Elasticity Index is obtained by ultrasonographic Shear Wave Elastography performed by two investigators on the same day. The inter- and intra-observer variation and day-to-day variation is calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Øre-Næse-Halsafdeling H, Aarhus University Hospital, Aarhus C, Denmark